CLINICAL TRIAL: NCT04376021
Title: The Effect of Physical Contact on Maternal Responsiveness and Breastfeeding Outcomes Among Low Income Mothers Participating in the California Border Healthy Start Program
Brief Title: Proyecto BEBE: The Effect of Babywearing Education on Breastfeeding Exclusivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurturely (Other)
Collaborators: Project Concern International (Other)
Responsible Party: Principal Investigator, Emily Little, Founder & Director, Nurturely
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 28
Record Dates: First submitted 2018-03-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Breastfeeding, Exclusive; Mother-Infant Interaction; Postpartum Depression
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Contact (Experimental): Baby carrier (and education) provided to mother to increase physical contact with baby
  Interventions: Behavioral: Babywearing
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Babywearing — Increase mother-infant physical contact through babywearing
  Arms: Physical Contact

SUMMARY:
To test the hypothesis that increased mother-infant physical contact affects the likelihood of mothers exclusively breastfeeding their child for the first six months of life, the investigators will randomly assign half of the participating mothers to receive a baby carrier to use with their baby (to facilitate increased physical contact) while the other half of babies and mothers will receive standard care.

DETAILED DESCRIPTION:
One hundred mothers participating in the California Border Healthy Start (CBHS) program will be randomly assigned to the physical contact group or the control group. Mothers in the physical contact group will be provided with an infant carrier to use from birth to facilitate increased mother-infant physical contact. In the control group, mothers will be provided with an infant carrier, but will not receive the carrier until postpartum week 24, once study measures have been collected. This type of multiple-baseline design will allow the investigators to objectively assess the effect of physical contact during the first six months, but will also ensure that mothers in both groups have the opportunity to benefit from the potentially positive intervention of a high quality infant carrier to promote increased mother-infant physical contact. The two groups will be compared on: 1) likelihood of exclusive breastfeeding, 2) extent of breastfeeding exclusivity (proportion of feeds that are breastmilk versus formula or other), 3) likelihood of initiating feeding in response to hunger cues versus crying (i.e., maternal responsiveness during feeding), 4) maternal score on the Edinburgh Postnatal Depression Scale (EPDS), 5) prevalence of breastfeeding difficulties, 6) score on the Mother-Infant Bonding Scale, and 7) beliefs about breastfeeding and infant care.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, participants:

* Must be a current participant in the CBHS program
* Must be 18 years of age or older
* Must be currently pregnant
* Must be fluent in either Spanish or English
* Must have consistent access to a smartphone with internet access (to fill out surveys and feeding logs)
* Must have a functioning email address Must be willing to share certain personal information with the researchers

Exclusion Criteria:

* Having a birth that does not result in a live, healthy, singleton infant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Proportion of infant feeds coming from breastmilk versus formula | Postpartum Week 24
  Self-report feeding log

SECONDARY OUTCOMES:
Score on Edinburgh Postnatal Depression Scale (EPDS) | Postpartum Week 6
  Standardized self-report questionnaire with a possible score from 0-30, with a higher score indicating increased depressive symptoms
Score on the Mother-Infant Bonding Questionnaire | Postpartum Week 24
  Standardized self-report questionnaire with a possible score from 0-30, with a higher score indicating increased problems with bonding
Score on the Proximal Care Beliefs Questionnaire | Postpartum Week 12
  Standardized self-report questionnaire with a possible score from 6-30, with a higher score indicating increased alignment with the caretaking practices of proximal care culture

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Little, PhD, Principal Investigator — Nurturely
Locations (1):
- Project Concern International, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Little EE, Bain L, Hahn-Holbrook J. Randomized controlled trial to prevent postpartum depressive symptomatology: An infant carrier intervention. J Affect Disord. 2023 Nov 1;340:871-876. doi: 10.1016/j.jad.2023.08.044. Epub 2023 Aug 15. PMID 37586649
- [Derived] Little EE, Cioffi CC, Bain L, Legare CH, Hahn-Holbrook J. An Infant Carrier Intervention and Breastfeeding Duration: A Randomized Controlled Trial. Pediatrics. 2021 Jul;148(1):e2020049717. doi: 10.1542/peds.2020-049717. Epub 2021 Jun 30. PMID 34193622